CLINICAL TRIAL: NCT05668910
Title: Development and Validation of a Blood-based Assay for Gastric Cancer Early Detection Using Multi-dimensional Analysis of Cell Free DNA Whole Methylome Sequencing-Protocol for an Observational, Case-control Study
Brief Title: Gastric Cancer Early Detection by Multi-dimensional Analysis of cfDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GeneCast Biotechnology Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Sponsor
Other Study IDs: D-P200110-MCCGW-HP-7-GC
Record Dates: First submitted 2022-12-12; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- malignant group: patients diagnosed with high grade Intraepithelial neoplasia or GC (> 50% of patients in stage I and II)
  Interventions: Genetic: whole genomic methylation and fragmentation profile analysis of cfDNA
- non-malignant group: healthy individuals and patients with non-atrophic gastritis, gastric ulcer, gastric polyp or other benign gastric diseases
  Interventions: Genetic: whole genomic methylation and fragmentation profile analysis of cfDNA

INTERVENTIONS:
Genetic: whole genomic methylation and fragmentation profile analysis of cfDNA — The assay for gastric cancer early detection will be built based on low-depth methylone sequencing followed with a multi-dimensional model construction with analysing several features such as methylation, fragmentation, and chromosomal copy number alternation.

SUMMARY:
To facilitate the early gastric cancer diagnosis, an assay based on assessing large-scale methylation and fragmentation profiles of the plasma cell free (cfDNA) will be developed and validated.

DETAILED DESCRIPTION:
Cancer-related features in cell-free DNA (cfDNA) fragments have gradually been identified and play essential roles for non-invasive early cancer detection. Integrated analysis of several cfDNA features have proven to achieve enhanced detection sensitivity as compared to single feature.

This study aims to develop and validate a novel blood-based whole methylome sequencing followed with a multi-dimensional model to analyze several features of cfDNA for GC early detection. Specifically, blood samples will be prospectively collected before gastroscopy. Cases and controls will be randomly divided into a training and a testing dataset at a ratio of 2:1. Plasma cfDNA will be isolated and extracted, followed with a bisulfite-free low-depth whole methylome sequencing. A multi-dimensional model named THorough Epigenetic Marker Integration Solution (THEMIS) including methylation, fragmentation, and chromosomal copy number alternation will be constructed in the training dataset. The performance of the model in differentiating cancer patients from non-cancer controls will then be evaluated in the testing dataset.

ELIGIBILITY:
Inclusion Criteria:

1. Complete clinical info;
2. Patients self-agree to join the study and with signed patient consent and good compliance.

The specific inclusion criteria for subjects to be included in the malignant group:

1. According to the definition of AJCC's 8th Edition Cancer Staging Manual, patients with gastric adenocarcinoma confirmed by histopathology and with pathological stages of stage I-IV, including patients with esophageal gastric junction adenocarcinoma (EGJ);
2. Has not previously received any local or systematic anti-tumor treatment.

Exclusion Criteria:

1. Diagnosed previously with any kind of malignant tumor;
2. Have received total or partial gastrectomy;
3. Have received bone marrow or organ transplantation;
4. Have received blood transfusion in the past 6 months;
5. Incomplete clinical info or unqualified to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll about 360 individuals who receive gastroscopy in The First Affiliated Hospital of Air Force Military Medical University (Xijing Hospital), Xi'an, Shaanxi province, China.
  Two groups will be formed based on gastroscopy results, malignant group and non-malignant group. The malignant group includes patients diagnosed with high grade Intraepithelial neoplasia or GC (> 50% of patients in stage I and II) while the non-malignant group contains healthy individuals and patients with non-atrophic gastritis, gastric ulcer, gastric polyp or other benign gastric diseases.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
The performance of each single feature and the ensemble model with integrated features for early GC detection | 18 months
  The efficacy of each single feature-based model and the ensemble model comparing with pathologic diagnostic results, the gold standard, and gastroscope diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).
The performance of each single feature and the ensemble model with integrated features for early GC detection in each clinical stage | 18 months
  The efficacy of each single feature-based model and the ensemble model comparing with pathologic diagnostic results, the gold standard, and gastroscope diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

SECONDARY OUTCOMES:
The performance of the ensemble model in combination of possible GC related biomarkers such as PG, G17, and/or Hp levels for early GC detection | 18 months
  The efficacy of the integrated model comparing with pathologic diagnostic results, the gold standard, and gastroscope diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Gang Ji, Principal Investigator — The First Affiliated Hospital of Air Force Military Medical University (Xijing Hospital), Xi'an, China
Locations (1):
- The First Affiliated Hospital of Air Force Military Medical University (Xijing Hospital), Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Han Y, Wei J, Wang W, Gao R, Shen N, Song X, Ni Y, Li Y, Xu LD, Chen W, Li X. Multidimensional Analysis of a Cell-Free DNA Whole Methylome Sequencing Assay for Early Detection of Gastric Cancer: Protocol for an Observational Case-Control Study. JMIR Res Protoc. 2023 Sep 20;12:e48247. doi: 10.2196/48247. PMID 37728978